CLINICAL TRIAL: NCT03612934
Title: The Influence of Specialist Palliative Care on the Exacerbation of Negative Symptoms, Life Quality and Performance Status of Patients With Advanced Breast Cancer
Brief Title: The Impact of SPC on Advanced Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Łukasz Pietrzyński, Principal Investigator, Silesian University of Medicine
Other Study IDs: SPC1
Record Dates: First submitted 2018-07-09; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Palliative Care; Quality of Life; Cancer, Breast
Keywords: Breast Cancer; palliative care; life quality; performance status; esas
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients under the age of 65 years: patients under the age of 65 years
  Interventions: Procedure: Specialist Palliative Care
- patients at the age of 65 years and over: patients at the age of 65 years and over
  Interventions: Procedure: Specialist Palliative Care

INTERVENTIONS:
Procedure: Specialist Palliative Care — In the research, Specialist Palliative Care was provided according to the guidelines established by Mid-Western Health Board in a Report of the National Advisory Committee on Palliative Care as well as according to recommendations of Polish Society of Palliative Medicine and Polish National Healthcare Fund. In order to ensure interdisciplinary and integrated palliative care, a team of specialists was appointed. Team members were engaged in the process of treatment of each patient during the time of the study and applied their specialist skills according to the needs of the patients

SUMMARY:
The aim of this prospective, observational study is the evaluation of the effectiveness of a 14-day Specialist Palliative Care therapy in participants with advanced breast cancer carried out in a stationary palliative care unit in Poland. The length of the entire study will be 36 months.

ELIGIBILITY:
Inclusion Criteria:

the patient's conscious consent for examination and the ability to fill in the form by the patient herself.

-

Exclusion Criteria:

* patients with cognitive disturbances disabling credible answers in the questionnaire, deceased patients or those discharged from the ward before 14 days of hospitalisation.

Ages: 33 Years to 91 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced stage breast cancer refered for a SPC treatment at palliative care department in Poland, Będzin.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Variation of intensification of patients negative symptoms before and after SPC | 14 days
  intensification of patients negative symptoms was assessed by Edmonton Symptom Assessment System (esas)
Variation of performance status of patients before and after SPC | 14 days
  performance status of patients was assessed by ECOG scale (Eastern Cooperative Oncology Group)
Variation of quality of life of patients before and after SPC | 14 days
  quality of life of patients of patients was assessed by quality of life uniscale (QoLU)

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga Jośko-Ochojska, prof, Study Chair — 4. Chair and Department of Medicine and Environmental Epidemiology Medical University of Silesia in Katowice; Łukasz Pietrzyńsi, Principal Investigator — 1. Medical University of Silesia, department of palliative medicine

IPD SHARING:
Plan to Share IPD: Undecided